CLINICAL TRIAL: NCT07109310
Title: A Prospective, Single-Center Clinical Validation Study of Transcri Ptomics-Based Biomarkers for Predicting Respiratory Infection Progression and Prognosis
Brief Title: A Validation Study on a Prognostic Prediction Model for Respiratory Tract Infections
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Xinlun Tian, Chief physician, professor, Peking Union Medical College Hospital
Other Study IDs: RTIModel-001
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Sepsis; Acute Respiratory Distress Syndrome; Community Acquired Pneumonia; Transcriptome
MeSH Terms: conditions — Sepsis; Respiratory Distress Syndrome; Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community-acquired pneumonia/sepsis group
  Interventions: Diagnostic Test: RTImodel001

INTERVENTIONS:
Diagnostic Test: RTImodel001 — This model was developed through transcriptome sequencing combined with machine learning to predict the risk of disease progression and clinical outcomes of respiratory tract infections

SUMMARY:
This study adopted a prospective, single-center, open-label design, aiming to evaluate the efficacy of the RTI clinical outcome prediction model in predicting clinical outcomes in subjects with acute respiratory tract infections.

In this study, the subjects were divided into the community-acquired pneumonia group and the sepsis group, including one baseline visit, one visit on the 7th day, and one visit on the 28th day.

During the research process, blood samples will be collected at the corresponding visiting points for the validation of the predictive model.

ELIGIBILITY:
Inclusion Criteria:

Community-acquired pneumonia group

* Age ≥18 years old;

  * Sign the informed consent form; ③ According to the researcher's judgment, be able to comply with the research visit; ④ Comply with the diagnostic criteria for community-acquired pneumonia in the Chinese Guidelines for the Diagnosis and Treatment of Community-Acquired Pneumonia in Adults (2016 Edition); ⑤ The time from onset to enrollment was ≤8 days. Sepsis Group
* Age ≥18 years old;

  * Sign the informed consent form; ③ According to the researcher's judgment, be able to comply with the research visit;

    * Patients who meets the sepsis 3.0 diagnostic criteria.

Exclusion Criteria:

Exclusion criteria

* Respiratory failure related to underlying heart and lung diseases;

  * Severe liver and kidney dysfunction, pregnancy or lactation period;

    * Meet the indications for organ transplantation or have undergone organ transplantation surgery in the past; ④ Known HIV infection; ⑤ Screening: Those who have experienced unstable angina pectoris or myocardial infarction within 30 days prior to the screening and have not received vascular recanalization treatment, as well as those with extensive cerebral hemorrhage; ⑥ Situations where researchers determine that enrollment is not appropriate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute respiratory tract infections
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Any of the following occurs: 1) Death; 2) Progress to sepsis (SOFA≥2 points); 3) Follow up for 28 days. | From enrollment to the end of follow-up at 28 days

SECONDARY OUTCOMES:
The changes of the seven-scale compared to the time of enrollment | From enrollment to the end of follow-up at 28 days
The changes in SOFA score compared to the time of enrollment. | From enrollment to the end of follow-up at 28 days

IPD SHARING:
Plan to Share IPD: No